CLINICAL TRIAL: NCT01727635
Title: The Long-term Effects of Body-mind-spirit Group Therapy on Close Relationships, Sleeping Quality, Depression, Quality of Life, Meaning of Life, and Saliva Cortisol Responses in Breast Cancer Survivors and Partners
Brief Title: The Long-term Effects of Body-mind-spirit Group Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200909010R
Record Dates: First submitted 2009-10-21; First posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Depression; Sleep
Keywords: Breast cancer, survivors, partners, group therapy
MeSH Terms: conditions — Depression; Breast Neoplasms | interventions — Psychotherapy, Group

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- counseling (Experimental): body-mind-spirit group therapy
  Interventions: Other: body-mind-spirit group therapy

INTERVENTIONS:
Other: body-mind-spirit group therapy — 8-session therapy
  Other Names: group therapy

SUMMARY:
Aims and objectives: This study aims to examine the effects of the body-mind-spirit group therapy on marital close relationships, sleeping quality, depression, quality of life, meaning of life, and salivary cortisol levels in metastatic breast cancer survivors and partners.

Methods: The design adopts the randomized controlled trial (RCT). The metastatic breast cancer survivors will be recruited from outpatient department of surgical at hospital. The partners will be invited to participate in this study through the survivors. The 120 dyad survivors and spouse will be randomly assigned into an experimental group or a control group. Survivors and spouse partners in an experimental group will receive 2 months time body-mind-spirit group therapy while those in a control will receive usual care in the same period of time. The outcome measures include Experiences in close relationships scale, Moss sleeping scale, Short-form 12 health-related quality of life questionnaires, Meaning of life questionnaire, BDI-II depression scale and salivary cortisol levels. Measurement time-points include pre intervention, post intervention (after 8 weekly group therapy), & then 3, 6, 12 months after the end of intervention for the maintenance effect. Univariate analyses will be performed to explore the basic characteristics of participants. The hierarchical linear model will be used to test the hypothesis the improvement is higher in intervention group than the control group in the effects of marital close relationships, sleeping quality, depression, meaning of life, quality of life, and salivary cortisol levels in metastatic breast cancer survivors and partners.

DETAILED DESCRIPTION:
Aims and objectives: This study aims to examine the effects of the body-mind-spirit group therapy on marital close relationships, sleeping quality, depression, quality of life, meaning of life, and salivary cortisol levels in metastatic breast cancer survivors and partners. Methods: The design adopts the randomized controlled trial (RCT). The metastatic breast cancer survivors will be recruited from outpatient department of surgical at hospital. The partners will be invited to participate in this study through the survivors. The 120 dyad survivors and spouse will be randomly assigned into an experimental group or a control group. Survivors and spouse partners in an experimental group will receive 2 months time body-mind-spirit group therapy while those in a control will receive usual care in the same period of time. The outcome measures include Experiences in close relationships scale, Moss sleeping scale, Short-form 12 health-related quality of life questionnaires, Meaning of life questionnaire, BDI-II depression scale and salivary cortisol levels. Measurement time-points include pre intervention, post intervention (after 8 weekly group therapy), & then 3, 6, 12 months after the end of intervention for the maintenance effect. Univariate analyses will be performed to explore the basic characteristics of participants. The hierarchical linear model will be used to test the hypothesis the improvement is higher in intervention group than the control group in the effects of marital close relationships, sleeping quality, depression, meaning of life, quality of life, and salivary cortisol levels in metastatic breast cancer survivors and partners.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of Survivors:

1. breast cancer patients who complete active treatments,
2. those who are willing to participate in the research,
3. those who currently do not receive any individual or group psychotherapy, AND
4. aged between 18 and 65.

Inclusion criteria of Spouse partners:

1. partners of breast cancer patient who complete active treatments,
2. those who are willing to participate in the research,
3. those who currently do not receive any individual or group psychotherapy, AND
4. aged between 18 and 65.

Exclusion Criteria:

Exclusion criteria of Survivors:

1. diagnosed as both breast cancer and other types of cancers,
2. those with adrenal function disorders (for example, Cushing syndrome, Addison's disease, adrenal tumor, pituitary tumor), OR
3. those who currently use antidepressants.

Exclusion criteria of Survivors:

1. diagnosed as adrenal function disorders (for example, Cushing syndrome, Addison's disease, adrenal tumor, pituitary tumor), OR
2. those who currently use antidepressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Diurnal Cortisol patterns | pre, post, 3months, 6months and 1year after end of treatment

SECONDARY OUTCOMES:
The Experiences in Close Relationships-Revised questionnaire | pre, post, 3months, 6months and 1year after end of treatment
Beck Depression Inventory | pre, post, 3months, 6months and 1year after end of treatment
Quality of life | pre, post, 3months, 6months and 1year after end of treatment
MOS sleep scale | pre, post, 3months, 6months and 1year after end of treatment
Meaning in Life Questionnaire | pre, post, 3months, 6months and 1year after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fei Hsiao, PhD, Principal Investigator — National Taiwan University
Locations (1):
- Department of Nursing, College of Medicine, National Taiwan University, Taipei, Taiwan